CLINICAL TRIAL: NCT05014581
Title: Preventing Cardiovascular Collapse With Vasopressors During Tracheal Intubation. The PREVENTION Randomized Multicenter Study
Brief Title: Preventing Cardiovascular Collapse With Vasopressors During Tracheal Intubation
Acronym: PREVENTION
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: University of Turin, Italy (Other)
Collaborators: Istituto Di Ricerche Farmacologiche Mario Negri (Other)
Responsible Party: Principal Investigator, Vincenzo Russotto, Principal Investigator, University of Turin, Italy
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PREVENTION
Record Dates: First submitted 2021-08-10; First posted 2021-08-20 (Actual); Last update posted 2025-03-28 (Actual); Status verified 2025-03

CONDITIONS: Critical Illness; Respiratory Failure
Keywords: tracheal intubation
MeSH Terms: conditions — Critical Illness; Respiratory Insufficiency | interventions — Norepinephrine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pre-emptive vasopressor (Experimental): Pre-emptive continuous infusion of norepinephrine during intubation
  Interventions: Drug: Noradrenaline
- No vasopressor (No Intervention): No pre-emptive administration of vasopressors

INTERVENTIONS:
Drug: Noradrenaline — Pre-emptive continuous infusion of noradrenaline during the peri-intubation period
  Other Names: Norepinephrine
  Arms: Pre-emptive vasopressor

SUMMARY:
Tracheal intubation (TI) is associated with a high risk of adverse events in critically ill patients and peri-intubation hemodynamic collapse is the most commonly observed. The primary aim of the PREVENTION trial is to compare the effect of the pre-emptive use of noradrenaline versus no peri-intubation use of noradrenaline on incidence of cardiovascular collapse following TI in adult critically ill patients. Patients with absolute indication or contraindication to vasopressor support will be excluded from this trial. Patients will be randomized 1:1 to a continuous infusion of noradrenaline started before induction titrated according to baseline mean arterial pressure. The primary outcome will be the incidence of cardiovascular collapse. Secondary outcomes will include lowest systolic blood pressure and cardiac arrest within 30 minutes from intubation.

DETAILED DESCRIPTION:
PREVENTION trial is a pragmatic, multi-center, un-blinded, parallel group, randomized study comparing the pre-emptive use of noradrenaline to no-vasopressors during the peri-intubation period of adult critically ill patients. Investigators hypothesize that the pre-emptive administration of noradrenaline would mitigate the incidence and severity of peri-intubation cardiovascular collapse. The study will include adult (18 yrs or older) critically ill patients needing in-hospital intubation, excluding patients with absolute indication or contraindication to vasopressors. Patients will be randomized to receive either a continuous infusion of noradrenaline started at least 8 minutes before induction vs no vasopressors during the peri-intubation period. All co-interventions will be provided according to clinician's judgement. The primary outcome of the study will be a composite of MAP < 60 mmHg or cardiac arrest. Secondary outcomes will include lowest systolic blood pressure < 30 minutes from induction, change in systolic blood pressure from baseline to the lowest value within 30 minutes from induction and cardiac arrest.

ELIGIBILITY:
Inclusion Criteria:

* Patient is admitted or scheduled for admission to a participating study hospital
* Planned procedure is tracheal intubation and planned operator is a provider expected to routinely perform endotracheal intubation in the participating unit
* Critical illness (i.e. life-threatening condition with intubation required for cardiorespiratory failure or neurological impairment)
* Administration of sedation (with or without neuromuscular blockade) is planned
* Age 18 years or older

Exclusion Criteria:

* No vasopressors/inotropes at the moment of screening for eligibility
* MAP < 60 mmHg or > 120 mmHg at the moment of screening for eligibility
* Urgency of intubation precludes safe performance of study procedures
* Intubation performed during cardiopulmonary resuscitation of a patient in cardiac arrest
* Enrolled in another clinical trial that is unapproved for co-enrollment
* Pregnant or suspected pregnancy

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 420 (Estimated)
Dates: Start 2024-08-01 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2026-04 (Estimated)

PRIMARY OUTCOMES:
Number of patients with cardiovascular collapse | 30 minutes from induction
  Composite outcome of mean arterial pressure < 60 mmHg or cardiac arrest

SECONDARY OUTCOMES:
Number of patients with cardiac arrest | 30 minutes from induction
  Development of either a shockable or non shockable rhythm associated with cardiac arrest
Number of patients with MAP < 60 mmHg | 30 minutes from induction
  Mean arterial pressure < 60 mmHg
Need for a rescue vasopressor | 30 minutes from induction
  Any unplanned administration of a vasopressor (either as bolus or continuous infusion)
Change in SBP value from last value before induction to lowest value | 30 minutes from induction
  Drop of the systolic blood pressure from baseline value to the lowest value registered by 30 minutes from induction
Lowest value of SBP | 30 minutes from induction
  Lowest systolic blood pressure
Number of patients with severe hypertension | 30 minutes from induction
  Mean arterial pressure > 120 mmHg

OTHER OUTCOMES:
Number of patients with cardiac arrhythmias | 30 minutes from induction
  Any ventricular or supraventricular arrhythmia
Number of patients with bradycardia | 30 minutes from induction
  Heart rate < 60 beats per minute
Signs of tissue/peripheral ischemia at noradrenaline infusion site | 24 hours
  Any sign of tissue/limb ischemia in case of peripheral vein infusion of noradrenaline
Need for new start of renal replacement therapy | 28 days from intubation
  Need to start either continuous or intermittent renal replacement therapy
Total amount of fluid administered (ml) | 30 minutes from induction
  Cumulative volume of fluids (ml)
First pass intubation success | 30 minutes from induction
  Confirmed intubation after a single attempt of laryngoscopy
Total amount of rescue vasopressors after induction | 30 minutes from induction
  Cumulative dose of any vasopressor administered either as a bolus or continuous infusion
ICU-free days | 28 days from intubation
  Total number of days outside the ICU up to 28 days
Ventilator-free days | 28 days from intubation
  Total number of days free from invasive mechanical ventilation
Vasopressor-free days | 28 days from intubation
  Total number of days free from any vasopressor administration
In-hospital mortality | 28 days from intubation
  Death during the hospital admission up to 28 days

CONTACTS AND LOCATIONS:
Overall Officials: Vincenzo Russotto, MD, Principal Investigator — University Hospital San Luigi Gonzaga; John G Laffey, MD, Study Chair — University Hospital Galway, NUI Galway, Ireland
Locations (6):
- CHU de Nantes, Nantes, France
- Galway University Hospitals, Galway, Ireland
- Italy (4):
  - Humanitas Research Hospital, Rozzano, Milan
  - University Hospital San Luigi Gonzaga, Orbassano, Turin
  - ASST Grande Ospedale Metropolitano Niguarda, Milan
  - Policlinico di Milano, Milan

REFERENCES:
- [Result] Russotto V, Myatra SN, Laffey JG, Tassistro E, Antolini L, Bauer P, Lascarrou JB, Szuldrzynski K, Camporota L, Pelosi P, Sorbello M, Higgs A, Greif R, Putensen C, Agvald-Ohman C, Chalkias A, Bokums K, Brewster D, Rossi E, Fumagalli R, Pesenti A, Foti G, Bellani G; INTUBE Study Investigators. Intubation Practices and Adverse Peri-intubation Events in Critically Ill Patients From 29 Countries. JAMA. 2021 Mar 23;325(12):1164-1172. doi: 10.1001/jama.2021.1727. PMID 33755076
- [Result] Russotto V, Myatra SN, Laffey JG. What's new in airway management of the critically ill. Intensive Care Med. 2019 Nov;45(11):1615-1618. doi: 10.1007/s00134-019-05757-0. Epub 2019 Sep 16. No abstract available. PMID 31529354
- [Result] Janz DR, Casey JD, Semler MW, Russell DW, Dargin J, Vonderhaar DJ, Dischert KM, West JR, Stempek S, Wozniak J, Caputo N, Heideman BE, Zouk AN, Gulati S, Stigler WS, Bentov I, Joffe AM, Rice TW; PrePARE Investigators; Pragmatic Critical Care Research Group. Effect of a fluid bolus on cardiovascular collapse among critically ill adults undergoing tracheal intubation (PrePARE): a randomised controlled trial. Lancet Respir Med. 2019 Dec;7(12):1039-1047. doi: 10.1016/S2213-2600(19)30246-2. Epub 2019 Oct 1. PMID 31585796